CLINICAL TRIAL: NCT01913405
Title: A Phase 3, Multi-Center, Open Label Study of Efficacy and Safety of PEGylated rFVIII (BAX 855) in Previously Treated Patients With Severe Hemophilia A Undergoing Surgical or Other Invasive Procedures
Brief Title: Phase 3 Efficacy and Safety Study of BAX 855 in Severe Hemophilia A Patients Undergoing Surgical Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 261204; 2013-001359-11 (EudraCT Number)
Record Dates: First submitted 2013-06-27; First posted 2013-08-01 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BAX855 (Experimental): Pre-operative loading dose: Single loading dose, pre-surgery administered based on each study participant's individual PK results as well as target trough level for type and character of surgery, dental or invasive procedure being performed. In general, major surgery will target an 80-150% FVIII trough level, and minor surgery will target an initial 30-100% FVIII trough level.
  Intra-operative and post-operative dosing of BAX855 must be based on pre-dosage measurements of FVIII and the type and character of the surgery performed.
  Interventions: Biological: PEGylated Recombinant factor VIII (rFVIII)

INTERVENTIONS:
Biological: PEGylated Recombinant factor VIII (rFVIII) — Lyophilized powder and solvent for solution for injection
  Other Names: BAX 855; ADYNOVATE

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of BAX 855 in severe hemophilia A previously treated (PTP) males, 12 to 65 years of age who are undergoing elective surgical or other invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participant requires an elective major or minor surgical, dental or other invasive procedure (e.g. biopsy, endoscopy).
* Participant and/or legal representative has/have provided signed informed consent.
* Participant has severe hemophilia A (Factor VIII (FVIII) level <1%) as confirmed by the central lab at screening or a documented FVIII activity level <1%.
* Participant was previously treated with FVIII concentrates with ≥150 documented exposure days (EDs).
* Participant is currently receiving prophylaxis or on-demand therapy with FVIII concentrate.
* Participant has a Karnofsky performance score of ≥60 at screening.
* Participant is human immunodeficiency virus negative (HIV-); or HIV+ with stable disease and CD4+ count ≥200 cells/mm^3, as confirmed by central laboratory at screening.
* Participant is Hepatitis C virus negative (HCV-) by antibody or PCR testing (if positive, antibody titer will be confirmed by PCR), as confirmed by central laboratory at screening; or HCV+ with chronic stable hepatitis as assessed by the investigator.
* Participant is willing and able to comply with the requirements of the study protocol.

Exclusion Criteria:

* Participant has detectable FVIII inhibitory antibodies (≥0.4 Bethesda Unit (BU) using the Nijmegen modification of the Bethesda assay) at screening as determined by the central laboratory or at any timepoint prior to screening (≥0.4 BU using the Nijmegen modification of the Bethesda assay or ≥0.6 BU using the Bethesda assay).
* History of ongoing or recent thrombotic disease, fibrinolysis or disseminated intravascular coagulation (DIC).
* Participant has a platelet count <100 x 10^9/L, as confirmed by central laboratory at screening.
* Participant has severe renal impairment (serum creatinine > 2.0 mg/dL), as confirmed by central laboratory at screening.
* Participant has severe chronic hepatic dysfunction (eg ≥5 X upper limit of normal alanine aminotransferase (ALT), as confirmed by the central laboratory at screening, or a documented International Normalized Ratio (INR) > 1.5).
* Participant has a known hypersensitivity towards mouse or hamster proteins, polysorbate 80 or to PEG.
* Participant is currently using or has recently (< 30 days) used pegylated drugs (other than BAX 855) prior to study participation or is scheduled to use such drugs during trial participation.
* Participant is currently participating in another clinical drug (other than BAX 855) or device study or use of another investigational product or device within 30 days prior to study entry.
* Participant has a diagnosis of an inherited or acquired hemostatic defect other than hemophilia A.
* Participant is currently receiving, or scheduled to receive during the course of the study, an immunomodulating drug (eg, systemic corticosteroid agent at a dose equivalent to hydrocortisone >10 mg/day, or alpha interferon) other than anti-retroviral chemotherapy.
* Participant has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect participant safety or compliance.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- United States (8):
  - University of Florida College of Medicine, Gainesville, Florida
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - University of Louisville, Louisville, Kentucky
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Bulgaria (2):
  - SHAT of Oncohaematology Diseases, Sofia
  - MHAT 'Sv. Marina', EAD, Varna
- Vilnius University Hospital Santariskiu Clinics, Public Institution, Vilnius, Lithuania
- Academisch Medisch Centrum, Amsterdam, Netherlands
- FSHI "Kirov SR Institute of Hematology and Blood Transfusion FMBA", Kirov, Russia
- Spain (4):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Regional Universitario de Malaga, Málaga, Málaga
  - Hospital Universitari i Politecnic La Fe, Valencia
- Universitaetsspital Zuerich, Zurich, Switzerland
- SI Institute of Blood Pathology and Transfusion Medicine of AMSU, Lviv, Ukraine
- United Kingdom (3):
  - Royal Free Hospital, London, Greater London
  - Great Ormond Street Hospital for Children, London, Greater London
  - Royal Manchester Children's Hospital, Manchester, Greater Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Brand B, Gruppo R, Wynn TT, Griskevicius L, Lopez Fernandez MF, Chapman M, Dvorak T, Pavlova BG, Abbuehl BE. Efficacy and safety of pegylated full-length recombinant factor VIII with extended half-life for perioperative haemostasis in haemophilia A patients. Haemophilia. 2016 Jul;22(4):e251-8. doi: 10.1111/hae.12963. Epub 2016 Jun 21. PMID 27328112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve study sites have enrolled participants in seven countries (US, Russia, UK, Bulgaria, Lithuania, Spain, Switzerland). There were 30 surgical enrollments in a total of 23 unique participants. Seven unique participants enrolled more than once, of whom five received study product for more than one surgical procedure.
Pre-assignment Details: A total of 23 participants provided informed consent and were screened for study participation. Of these, 22 unique participants (29 surgical enrollments) were exposed to study product. One participant discontinued prior to surgery and one subject discontinued after surgery.
Groups:
- BAX855: Pre-operative loading dose: Single loading dose, pre-surgery administered based on each study participant's individual PK results as well as target trough level for type and nature of surgery, dental or invasive procedure being performed. In general, major surgery will target an 80-100% FVIII trough level, and minor surgery will target an initial 30-60% FVIII trough level. Intra-operative and post-operative dosing of BAX855 must be based on pre-dosage measurements of FVIII and the type and nature of the surgery performed.
Period: Overall Study
Arm/Group | BAX855
Started | 22
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | BAX855
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Global Hemostatic Efficacy Assessment Score (GHEA) - Composed of 3 Individual Ratings
Description: GHEA=Sum of 1-3 ratings: Excellent: 7-9 (no category <2), Good: 5-7 (no category <1), Fair: 3-4 (no category <1) 1. Intraoperative and 2. Postoperative (postoperative day 1) hemostatic efficacy assessments: Excellent=3: Blood Loss (BL) ≤ than expected for procedure type in non-hemophilic population (NHP) (≤100%), Good=2: BL ≤50% more than expect. for procedure type in NHP (101-150%), Fair=1: BL >50% more than expect. for procedure type in NHP (>150%), None=0: Significant bleeding-requiring rescue therapy (RT) 3. Perioperative hemostatic efficacy assessment (day 14 or discharge, whatever is first): Excellent=3: BL and required blood transfusions (BT) less than or similar (≤100%) to that expected for procedure type in NHP, Good=2: BL ≤50% more (101-150%) and BT less than or similar to that expected for procedure type in NHP, Fair=1: BL >50% more (>150%) and BT greater than expected in NHP, None=0: Significant bleeding-requiring RT, BT substantially greater than expected in NHP
Time Frame: Hemostatic efficacy assessments were performed intraoperatively, postoperatively on day 1 (approximately 24 hours after surgery) and perioperatively at day 14 or discharge (whichever was first).
Population: Full analysis group comprises groups major orthopedic and non-orthopedic and minor surgery. Main analysis was done on the full analysis group (at least one hemostatic assessment available) and supportive analysis was done on the per protocol analysis group (all hemostatic assessments available).
Measure: Number (90% Confidence Interval); unit: Percentage of surgeries
Units Other Than Participants: Surgeries
Groups:
- Full Analysis Group: All participants treated with BAX855 with available GHEA score.
- Major Orthopedic Surgery: All participants treated with BAX855 for major orthopedic surgery.
- Major Non-orthopedic Surgery: All participants treated with BAX855 for major non-orthopedic surgery.
- Minor Surgery: All participants treated with BAX855 for minor surgery.
- Per Protocol Analysis Group: All participants treated with BAX855 with all 3 hemostatic efficacy assessments available. Only subjects who met all study entry criteria and who had no major protocol violation that impacted hemostatic efficacy assessment were included in this group.
Arm/Group | Full Analysis Group | Major Orthopedic Surgery | Major Non-orthopedic Surgery | Minor Surgery | Per Protocol Analysis Group
Number analyzed (Participants) | 20 | 12 | 6 | 3 | 11
Number analyzed (Surgeries) | 24 | 14 | 7 | 3 | 12
Percentage of surgeries
  Treatment success (GHEA score excellent or good) | 100.0 [88.3 to 100.0] | 100.0 [80.7 to 100.0] | 100.0 [65.2 to 100.0] | 100.0 [36.8 to 100.0] | 100.0 [77.9 to 100.0]
  Excellent | 100.0 [88.3 to 100.0] | 100.0 [80.7 to 100.0] | 100.0 [65.2 to 100.0] | 100.0 [36.8 to 100.0] | 100.0 [77.9 to 100.0]
  Good | 0.0 [0.0 to 11.7] | 0.0 [0.0 to 19.3] | 0.0 [0.0 to 34.8] | 0.0 [0.0 to 63.2] | 0.0 [0.0 to 22.1]

2. Secondary Outcome: Intraoperative Blood Loss
Description: Actual intraoperative blood loss was assessed at the end of surgery and was compared to the estimated volume of expected average and maximum blood loss in a hemostatically normal individual of the same sex, age and stature as the study participant. Expected intraoperative blood loss was predicted preoperatively by the investigator/surgeon.
Time Frame: From initiation of surgery until end of surgery.
Population: The full analysis group comprises the groups with major orthopedic, major non-orthopedic and minor surgery.
Measure: Median (Inter-Quartile Range); unit: Milliliter
Units Other Than Participants: Surgeries
Groups:
- Full Analysis Group: All participants treated with BAX855 with at least one available hemostatic assessment.
Arm/Group | Full Analysis Group | Major Orthopedic Surgery | Major Non-orthopedic Surgery | Minor Surgery
Number analyzed (Participants) | 21 | 12 | 6 | 4
Number analyzed (Surgeries) | 26 | 14 | 7 | 5
Milliliter
  Actual blood loss: number analyzed (Participants) | 20 | 12 | 5 | 4
  Actual blood loss: number analyzed (Surgeries) | 25 | 14 | 6 | 5
  Actual blood loss | 10 [4 to 30] | 10 [10 to 30] | 4.5 [3 to 50] | 5 [0 to 15]
  Predicted average blood loss | 20 [5 to 150] | 150 [10 to 150] | 10 [5 to 50] | 5 [0 to 15]
  Difference from predicted average blood loss: number analyzed (Participants) | 20 | 12 | 5 | 4
  Difference from predicted average blood loss: number analyzed (Surgeries) | 25 | 14 | 6 | 5
  Difference from predicted average blood loss | 6 [0 to 135] | 125 [0 to 140] | 1.5 [0 to 6] | 0 [0 to 0]
  Predicted maximum blood loss | 100 [7 to 300] | 300 [100 to 300] | 20 [5 to 150] | 5 [0 to 30]
  Difference from predicted maximum blood loss: number analyzed (Participants) | 20 | 12 | 5 | 4
  Difference from predicted maximum blood loss: number analyzed (Surgeries) | 25 | 14 | 6 | 5
  Difference from predicted maximum blood loss | 100 [4 to 280] | 275 [95 to 290] | 25 [3 to 100] | 0 [0 to 15]

3. Secondary Outcome: Postoperative Blood Loss
Description: Actual post-operative blood loss assessed at postoperative day 1 was compared to the estimated volume of expected average and maximum blood loss in a hemostatically normal individual of the same sex, age and stature as the study participant. Expected postoperative blood loss was predicted pre-operatively by the investigator/surgeon.
Time Frame: From completion of surgery until 24 hours after surgery.
Population: The full analysis group comprises the groups with major orthopedic, major non-orthopedic and minor surgery.
Measure: Median (Inter-Quartile Range); unit: Milliliter
Units Other Than Participants: Surgeries
Arm/Group | Full Analysis Group | Major Orthopedic Surgery | Major Non-orthopedic Surgery | Minor Surgery
Number analyzed (Participants) | 21 | 12 | 6 | 4
Number analyzed (Surgeries) | 26 | 14 | 7 | 5
Milliliter
  Actual blood loss: number analyzed (Participants) | 13 | 7 | 4 | 3
  Actual blood loss: number analyzed (Surgeries) | 16 | 9 | 4 | 3
  Actual blood loss | 10 [0 to 825] | 750 [15 to 1100] | 1 [0 to 33.5] | 0 [0 to 4]
  Predicted average blood loss | 27.5 [0 to 300] | 213.5 [30 to 700] | 1 [0 to 25] | 0 [0 to 0]
  Difference from predicted average blood loss: number analyzed (Participants) | 13 | 7 | 4 | 3
  Difference from predicted average blood loss: number analyzed (Surgeries) | 16 | 9 | 4 | 3
  Difference from predicted average blood loss | -7.5 [-125 to 4] | -50 [-400 to -15] | 4 [-7.5 to 16.5] | 0 [0 to 196]
  Predicted maximum blood loss | 75 [0 to 600] | 450 [100 to 1200] | 2 [0 to 50] | 0 [0 to 0]
  Difference from predicted maximum blood loss: number analyzed (Participants) | 13 | 7 | 4 | 3
  Difference from predicted maximum blood loss: number analyzed (Surgeries) | 16 | 9 | 4 | 3
  Difference from predicted maximum blood loss | 67.5 [0 to 148] | 100 [0 to 300] | 34 [9 to 67.5] | 0 [0 to 196]

4. Secondary Outcome: Overall Perioperative Blood Loss
Description: Actual overall perioperative blood loss (assessed at the end of surgery, at postoperative day 1 and until discharge or day 14 - whichever is first) was compared to the estimated volume of expected average and maximum blood loss in a hemostatically normal individual of the same sex, age and stature as the study participant. Expected perioperative blood loss was predicted pre-operatively by the investigator/surgeon.
Time Frame: From start of surgery until discharge or day 14, whichever occurred first.
Population: The full analysis group comprises the groups with major orthopedic, major non-orthopedic and minor surgery.
Measure: Median (Inter-Quartile Range); unit: Milliliter
Units Other Than Participants: Surgeries
Arm/Group | Full Analysis Group | Major Orthopedic Surgery | Major Non-orthopedic Surgery | Minor Surgery
Number analyzed (Participants) | 21 | 12 | 6 | 4
Number analyzed (Surgeries) | 26 | 14 | 7 | 5
Milliliter
  Actual blood loss: number analyzed (Participants) | 20 | 12 | 5 | 4
  Actual blood loss: number analyzed (Surgeries) | 25 | 14 | 6 | 5
  Actual blood loss | 50 [5 to 305] | 246 [15 to 1210] | 5.5 [3 to 50] | 9 [0 to 15]
  Predicted average blood loss | 40 [5 to 800] | 675 [30 to 1000] | 20 [5 to 50] | 0 [0 to 15]
  Difference from predicted average blood loss: number analyzed (Participants) | 20 | 12 | 5 | 4
  Difference from predicted average blood loss: number analyzed (Surgeries) | 25 | 14 | 6 | 5
  Difference from predicted average blood loss | 0 [-50 to 20] | -5 [-210 to 25] | 2.5 [0 to 14] | 0 [0 to 0]
  Predicted maximum blood loss | 125 [20 to 1500] | 1500 [100 to 1500] | 20 [6 to 150] | 0 [0 to 30]
  Difference from predicted maximum blood loss: number analyzed (Participants) | 20 | 12 | 5 | 4
  Difference from predicted maximum blood loss: number analyzed (Surgeries) | 25 | 14 | 6 | 5
  Difference from predicted maximum blood loss | 64 [6 to 250] | 122.5 [50 to 400] | 5.5 [0 to 64] | 0 [0 to 15]

5. Secondary Outcome: Transfusion Requirements
Description: Volume of blood, red blood cells, platelets, and other blood products transfused. Only packed red blood cells were transfused in this study.
Time Frame: From initiation of the surgery to 24 hours after completion of the surgery.
Population: The full analysis group comprises the groups with major orthopedic, major non-orthopedic and minor surgery. Only participants who received blood transfusions are included in this analysis.
Measure: Mean (Standard Deviation); unit: Milliliter
Units Other Than Participants: Surgeries
Arm/Group | Full Analysis Group | Major Orthopedic Surgery | Major Non-orthopedic Surgery | Minor Surgery
Number analyzed (Participants) | 3 | 2 | 1 | 0
Number analyzed (Surgeries) | 4 | 3 | 1 | 0
Milliliter | 438.0 (152.86) | 384.0 (132.49) | 600.0 (NA) — only 1 participant analyzed |

6. Secondary Outcome: Occurrence of Bleeding Episodes and Additional Need for Surgical Intervention
Description: Any clinically relevant bleeding episodes (as assessed by the investigator) as well as the need for any further surgical interventions were recorded. If the subject had not resumed his previous treatment after discharge, the occurrence and treatment of bleeding episodes were recorded in the subject's diary.
Time Frame: Intra- and post-operative period, until the last intensified treatment after hospital discharge (minor surgery 1-3 days, major surgery average approximately 2 weeks)
Population: Only surgeries/participants that have encountered bleeding episodes are reported for the analysis of bleeding episodes (5 surgeries in 5 participants) and all surgeries/participants are reported for the analysis of the need for surgical intervention.
Measure: Number; unit: Events
Units Other Than Participants: Surgeries
Arm/Group | Full Analysis Group | Major Orthopedic Surgery | Major Non-orthopedic Surgery | Minor Surgery
Number analyzed (Participants) | 21 | 12 | 6 | 4
Number analyzed (Surgeries) | 26 | 14 | 7 | 5
Events
  Bleeding episodes site mucosal: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes site mucosal: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes site mucosal | 2 | 0 | 1 | 1
  Bleeding episodes site joint: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes site joint: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes site joint | 1 | 1 | 0 | 0
  Bleeding episodes site gastrointestinal: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes site gastrointestinal: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes site gastrointestinal | 1 | 0 | 1 | 0
  Bleeding episodes site muscle: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes site muscle: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes site muscle | 1 | 1 | 0 | 0
  Bleeding episodes cause spontaneous: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes cause spontaneous: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes cause spontaneous | 0 | 0 | 0 | 0
  Bleeding episodes cause inury: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes cause inury: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes cause inury | 5 | 2 | 2 | 1
  Bleeding episodes severity mild: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes severity mild: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes severity mild | 3 | 1 | 1 | 1
  Bleeding episodes severity moderate: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes severity moderate: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes severity moderate | 1 | 0 | 1 | 0
  Bleeding episodes severity severe: number analyzed (Participants) | 5 | 2 | 2 | 1
  Bleeding episodes severity severe: number analyzed (Surgeries) | 5 | 2 | 2 | 1
  Bleeding episodes severity severe | 1 | 1 | 0 | 0
  Additional need for surgery | 0 | 0 | 0 | 0

7. Secondary Outcome: Consumption of BAX855
Description: Daily and total weight-adjusted consumption of BAX855 per subject.
Time Frame: From initial loading dose until discharge for daily weight-adjusted dose and from first infusion (PK/IR) until end of study for total weight-adjusted dose.
Population: The full analysis group comprises the groups with major orthopedic, major non-orthopedic and minor surgery. Number of surgeries/participants with BAX855 consumption varies on each postoperative day.
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Surgeries
Arm/Group | Full Analysis Group | Major Orthopedic Surgery | Major Non-orthopedic Surgery | Minor Surgery
Number analyzed (Participants) | 21 | 12 | 6 | 4
Number analyzed (Surgeries) | 26 | 14 | 7 | 5
IU/kg
  Total weight adjusted BAX855 consumption | 562.076 (343.7305) | 746.103 (320.4581) | 507.881 (161.8075) | 122.673 (20.0076)
  Preoperative | 62.492 (15.7678) | 69.442 (14.4532) | 56.852 (14.8899) | 50.928 (12.2700)
  Postoperative Day 0: number analyzed (Participants) | 14 | 9 | 5 | 1
  Postoperative Day 0: number analyzed (Surgeries) | 18 | 11 | 6 | 1
  Postoperative Day 0 | 34.195 (13.6755) | 37.082 (16.0160) | 31.141 (7.5641) | 20.762 (NA) — Standard deviation not calculated as only 1 surgery analyzed
  Postoperative Day 1: number analyzed (Participants) | 20 | 12 | 6 | 3
  Postoperative Day 1: number analyzed (Surgeries) | 24 | 14 | 6 | 4
  Postoperative Day 1 | 56.409 (24.8718) | 62.005 (25.4147) | 50.698 (29.2373) | 45.388 (12.0692)
  Postoperative Day 2: number analyzed (Participants) | 16 | 11 | 6 | 0
  Postoperative Day 2: number analyzed (Surgeries) | 19 | 13 | 6 | 0
  Postoperative Day 2 | 51.697 (27.7558) | 52.445 (27.4771) | 50.076 (30.9322) |
  Postoperative Day 3: number analyzed (Participants) | 14 | 10 | 5 | 0
  Postoperative Day 3: number analyzed (Surgeries) | 17 | 12 | 5 | 0
  Postoperative Day 3 | 45.023 (24.2793) | 47.139 (27.1069) | 39.943 (17.0764) |
  Postoperative Day 4: number analyzed (Participants) | 13 | 10 | 4 | 0
  Postoperative Day 4: number analyzed (Surgeries) | 16 | 12 | 4 | 0
  Postoperative Day 4 | 36.593 (12.2194) | 38.009 (13.6782) | 32.345 (5.3374) |
  Postoperative Day 5: number analyzed (Participants) | 9 | 8 | 2 | 0
  Postoperative Day 5: number analyzed (Surgeries) | 12 | 10 | 2 | 0
  Postoperative Day 5 | 32.240 (15.1497) | 32.333 (15.1071) | 31.775 (21.6822) |
  Postoperative Day 6: number analyzed (Participants) | 7 | 6 | 2 | 0
  Postoperative Day 6: number analyzed (Surgeries) | 9 | 7 | 2 | 0
  Postoperative Day 6 | 34.135 (13.3132) | 35.198 (12.8578) | 30.415 (19.7589) |
  Postoperative Day 7: number analyzed (Participants) | 4 | 3 | 1 | 0
  Postoperative Day 7: number analyzed (Surgeries) | 4 | 3 | 1 | 0
  Postoperative Day 7 | 22.955 (6.0531) | 24.866 (5.7495) | 17.223 (NA) — Standard deviation not calculated as only 1 surgery analyzed |
  Postoperative Day 8+: number analyzed (Participants) | 2 | 2 | 0 | 0
  Postoperative Day 8+: number analyzed (Surgeries) | 2 | 2 | 0 | 0
  Postoperative Day 8+ | 136.808 (139.3781) | 136.808 (139.3781) |  |

8. Secondary Outcome: Pharmacokinetics (PK) - Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-∞)
Description: Following at least a 72 hour washout period a single dose of BAX855 was administered. The PK profiles was used to guide dosing and dosing frequency during the perioperative time period. The area under the plasma concentration/time curve from time 0 to infinity (AUC 0-inf) and the area under the first movement curve from time 0 to infinity (AUMC 0-inf) was calculated as the sum of AUC and AUMC from time 0 to the time of the last quantifiable concentration plus a tail area correction calculated as Ct/λz and Ct/λz(t+1/λz), respectively, where Ct is the last quantifiable concentration, t is the time of last quantifiable concentration and λz is the terminal or disposition rate constant. Main analysis was done on the one-stage clotting assay results, supportive analysis was done on the chromogenic assay results.
Time Frame: PK measurements were done within 30 minutes pre-infusion, and post infusion at 15 (± 5) minutes, 3 hours (± 30 minutes), 9 hours (± 30 minutes), 32 (± 2) hours, 56 (± 4) hours and 96 (± 4) hours.
Measure: Mean (Standard Deviation); unit: IU*h/dL
Units Other Than Participants: Surgeries
Groups:
- Pharmacokinetic Analysis Group: All participants who underwent a pharmacokinetic assessment with BAX855 infusion.
Arm/Group | Pharmacokinetic Analysis Group
Number analyzed (Participants) | 20
Number analyzed (Surgeries) | 25
IU*h/dL
  One-stage clotting assay | 2743.3 (751.83)
  Chromogenic assay | 3201.8 (1019.13)

9. Secondary Outcome: Pharmacokinetics (PK) - Area Under the Plasma Concentration/Time Curve From Time 0 to 96 Hours Post-infusion (AUC0-96h)
Description: Following at least a 72 hour (h) washout period a single dose of BAX855 will be administered. The PK profiles was used to guide dosing and dosing frequency during the perioperative time period. The area under the plasma concentration/time curve from time 0 to 96 hours postinfusion (AUC 0-96h) was computed using the linear trapezoidal rule. For the calculation of AUC 0-96h the levels at 96 hours were linearly interpolated/extrapolated from the 2 nearest sampling time points. Main analysis was done on the one-stage clotting assay results, supportive analysis was done on the chromogenic assay results.
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: IU*h/dL
Units Other Than Participants: Surgeries
Groups:
- Pharmocokinetic Analysis Group: All participants who underwent a pharmacokinetic assessment with BAX855 infusion.
Arm/Group | Pharmocokinetic Analysis Group
Number analyzed (Participants) | 20
Number analyzed (Surgeries) | 25
IU*h/dL
  One-stage clotting assay | 2701.3 (719.52)
  Chromogenic assay | 3153.7 (980.27)

10. Secondary Outcome: Pharmacokinetics (PK) - Terminal Half-life (T1/2)
Description: Following at least a 72 hour washout period a single dose of BAX855 will be administered. The PK profiles will be used to guide dosing and dosing frequency during the perioperative time period. Terminal or disposition half-life (HL) was calculated as log e(2)/λz where the terminal or disposition rate constant (λz) was estimated as the slope of a log-linear least squares regression model. Main analysis was done on the one-stage clotting assay results, supportive analysis was done on the chromogenic assay results. Terminal half life is the time it takes for the plasma concentration or the amount of drug in the body to be reduced by 50%.
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: Hours
Units Other Than Participants: Surgeries
Arm/Group | Pharmacokinetic Analysis Group
Number analyzed (Participants) | 20
Number analyzed (Surgeries) | 25
Hours
  One-stage clotting assay | 14.63 (3.179)
  Chromogenic assay | 14.53 (3.137)

11. Secondary Outcome: Pharmacokinetics (PK) - Mean Residence Time (MRT)
Description: Following at least a 72 hour washout period a single dose of BAX855 will be administered. The PK profiles will be used to guide dosing and dosing frequency during the perioperative time period. Mean residence time (MRT) was calculated as total area under the moment curve divided by the total area under the curve. Main analysis was done on the one-stage clotting assay results, supportive analysis was done on the chromogenic assay results.
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: Hours
Units Other Than Participants: Surgeries
Arm/Group | Pharmacokinetic Analysis Group
Number analyzed (Participants) | 20
Number analyzed (Surgeries) | 25
Hours
  One-stage clotting assay | 19.26 (4.901)
  Chromogenic assay | 18.68 (4.160)

12. Secondary Outcome: Pharmacokinetics (PK) - Clearance (CL)
Description: Following a 72 hour washout period a single dose of BAX855 will be administered. The PK profiles will be used to guide dosing and dosing frequency during the perioperative time period. Systemic clearance (CL) was calculated as the dose in IU/kg divided by the total AUC. Main analysis was done on the one-stage clotting assay results, supportive analysis was done on the chromogenic assay results. h = hours
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: dL/(kg*h)
Units Other Than Participants: Surgeries
Arm/Group | Pharmacokinetic Analysis Group
Number analyzed (Participants) | 20
Number analyzed (Surgeries) | 25
dL/(kg*h)
  One-stage clotting assay | 0.02347 (0.006821)
  Chromogenic assay | 0.02042 (0.006041)

13. Secondary Outcome: Pharmacokinetics (PK) - Apparent Volume of Distribution at Steady State (Vss)
Description: Following at least a 72 hour washout period a single dose of BAX855 will be administered. The PK profiles will be used to guide dosing and dosing frequency during the perioperative time period. Apparent steady state volume of distribution (Vss) was calculated as dose multiplied with AUMC(0-inf) divided by AUC(0-inf) to square. Main analysis was done on the one-stage clotting assay results, supportive analysis was done on the chromogenic assay results.
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: dL/kg
Units Other Than Participants: Surgeries
Arm/Group | Pharmacokinetic Analysis Group
Number analyzed (Participants) | 20
Number analyzed (Surgeries) | 25
dL/kg
  One-stage clotting assay | 0.4316 (0.09633)
  Chromogenic assay | 0.3673 (0.09559)

14. Secondary Outcome: Pharmacokinetics (PK) - Incremental Recovery(IR)
Description: Following at least a 72 hour washout period a single dose of BAX855 will be administered. The PK profiles will be used to guide dosing and dosing frequency during the perioperative time period. Incremental recovery (IR) was calculated as C post infusion minus C pre-infusion divided by the dose. Main analysis was done on the one-stage clotting assay results, supportive analysis was done on the chromogenic assay results.
Time Frame: as for outcome 8
Population: For measurement at 15 min post-infusion only 23 surgeries in 18 participants were available for analysis.
Measure: Mean (Standard Deviation); unit: (IU/dL):(IU/kg)
Units Other Than Participants: Surgeries
Arm/Group | Pharmacokinetic Analysis Group
Number analyzed (Participants) | 20
Number analyzed (Surgeries) | 25
(IU/dL):(IU/kg)
  IR at 15 min post infusion - one-stage clotting: number analyzed (Participants) | 18
  IR at 15 min post infusion - one-stage clotting: number analyzed (Surgeries) | 23
  IR at 15 min post infusion - one-stage clotting | 2.106 (0.3823)
  IR at 15 min post infusion - chromogenic: number analyzed (Participants) | 18
  IR at 15 min post infusion - chromogenic: number analyzed (Surgeries) | 23
  IR at 15 min post infusion - chromogenic | 2.721 (0.5981)
  IR at Cmax - one-stage clotting | 2.123 (0.4041)
  IR at Cmax - chromogenic | 2.677 (0.5960)

15. Secondary Outcome: Development of Inhibitory Antibodies to Factor VIII (FVIII)
Description: Immunogenicity assessment using FVIII inhibitor by Nijmegen method. A 72-hour washout period is required prior to immunogenicity tests.
Time Frame: Up to 105 days prior to surgery (Screening visit); and End of Study Visit (variable for each participant and depends on the nature of the invasive procedure (treatment period ranged from 43 days to 162 days).
Population: The safety analysis data set was used for the analysis of this outcome measure including all participants who received at least one infusion of BAX855.
Measure: Count of Participants; unit: Participants
Arm/Group | BAX855
Number analyzed (Participants) | 22
Participants | 0

16. Secondary Outcome: Development of Treatment Emerging Binding Antibodies to Factor VIII (FVIII), Treatment Emergent Binding Antibodies to PEGylated Recombinant FVIII (BX855), and Treatment Emerging Binding Antibodies to Polyethylene Glycol (PEG)
Description: A 72-hour washout period is required prior to immunogenicity tests.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | BAX855
Number analyzed (Participants) | 22
Participants
  Treatment emerging binding antibodies to FVIII IgG | 0
  Treatment emerging binding antibodies to FVIII IgM | 0
  Treatment emerging binding antibodies to BAX855IgG | 0
  Treatment emerging binding antibodies to BAX855IgM | 0
  Treatment emerging binding antibodies to PEG IgG | 0
  Treatment emerging binding antibodies to PEG IgM | 0

17. Secondary Outcome: Development of Treatment Emerging Anti-chinese Hamster Ovary (CHO) Antibodies
Description: A 72-hour washout period is required prior to immunogenicity tests.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | BAX855
Number analyzed (Participants) | 22
Participants | 0

18. Secondary Outcome: Occurrence of Thrombotic Events
Time Frame: Throughout the entire study period from screening to completion/termination. For each participant the duration of treatment and the entire study period depended on the nature of the invasive procedure (ranged from 43 days to 162 days).
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | BAX855
Number analyzed (Participants) | 22
Participants | 0

19. Secondary Outcome: Incidence of Severe Allergic Reactions (e.g. Anaphylaxis)
Time Frame: as for outcome 18
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | BAX855
Number analyzed (Participants) | 22
Participants | 0

20. Secondary Outcome: Other Investigational Product (IP) - Related Adverse Events
Time Frame: as for outcome 18
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | BAX855
Number analyzed (Participants) | 22
Participants | 2

21. Secondary Outcome: Clinically Significant Changes in Vital Signs - Body Temperature
Description: Changes in body temperature were assessed 15 minutes after the PK/IR infusion and compared to the pre-infusion values.
Time Frame: Vital signs measurement prior to the PK/IR infusion and 15 minutes post-infusion.
Population: The safety analysis data set was used for the analysis of this outcome measure including all participants who received at least one infusion of BAX855. Pre-infusion and 15 min post-infusion vital signs measurements are not available for all surgeries. 15 min. post-infusion measure includes 1 hour post infusion measure for 2 subjects.
Measure: Median (Inter-Quartile Range); unit: °Celsius
Units Other Than Participants: Surgeries
Arm/Group | BAX855
Number analyzed (Participants) | 22
Number analyzed (Surgeries) | 29
°Celsius
  Pre-infusion: number analyzed (Participants) | 20
  Pre-infusion: number analyzed (Surgeries) | 25
  Pre-infusion | 36.60 [36.30 to 36.70]
  15 minutes post infusion: number analyzed (Participants) | 19
  15 minutes post infusion: number analyzed (Surgeries) | 23
  15 minutes post infusion | 36.60 [36.20 to 36.70]
  Change at 15 minutes post infusion: number analyzed (Participants) | 19
  Change at 15 minutes post infusion: number analyzed (Surgeries) | 23
  Change at 15 minutes post infusion | 0.00 [-0.10 to 0.20]

22. Secondary Outcome: Clinically Significant Changes in Vital Signs - Systolic and Diastolic Blood Pressure (BP)
Description: Changes in systolic and diastolic blood pressure (mmHg) were assessed 15 minutes after the PK/IR infusion and compared to the pre-infusion values.
Time Frame: Vital signs measurement prior to the PK/IR infusion and 15 minutes post-infusion.
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: mmHg
Units Other Than Participants: Surgeries
Arm/Group | BAX855
Number analyzed (Participants) | 22
Number analyzed (Surgeries) | 29
mmHg
  Systolic BP: Pre-infusion: number analyzed (Participants) | 20
  Systolic BP: Pre-infusion: number analyzed (Surgeries) | 25
  Systolic BP: Pre-infusion | 120 [115.0 to 125.0]
  Systolic BP: 15 minutes post infusion: number analyzed (Participants) | 19
  Systolic BP: 15 minutes post infusion: number analyzed (Surgeries) | 23
  Systolic BP: 15 minutes post infusion | 115.0 [110.0 to 125.0]
  Systolic BP: Change at 15 minutes post infusion: number analyzed (Participants) | 19
  Systolic BP: Change at 15 minutes post infusion: number analyzed (Surgeries) | 23
  Systolic BP: Change at 15 minutes post infusion | -5.0 [-5.0 to 4.0]
  Diastolic BP: Pre-infusion: number analyzed (Participants) | 20
  Diastolic BP: Pre-infusion: number analyzed (Surgeries) | 25
  Diastolic BP: Pre-infusion | 75.0 [69.0 to 80.0]
  Diastolic BP: 15 minutes post infusion: number analyzed (Participants) | 19
  Diastolic BP: 15 minutes post infusion: number analyzed (Surgeries) | 23
  Diastolic BP: 15 minutes post infusion | 75.0 [70.0 to 80.0]
  Diastolic BP: Change at 15 minutes post infusion: number analyzed (Participants) | 19
  Diastolic BP: Change at 15 minutes post infusion: number analyzed (Surgeries) | 23
  Diastolic BP: Change at 15 minutes post infusion | 0.0 [-5.0 to 1.0]

23. Secondary Outcome: Clinically Significant Changes in Vital Signs - Respiratory Rate
Description: Changes in Respiratory rate were assessed 15 minutes after the PK/IR infusion and compared to the pre-infusion values.
Time Frame: Vital signs measurement prior to the PK/IR infusion and 15 minutes post-infusion.
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: breaths/minute
Units Other Than Participants: Surgeries
Arm/Group | BAX855
Number analyzed (Participants) | 22
Number analyzed (Surgeries) | 29
breaths/minute
  Pre-infusion: number analyzed (Participants) | 20
  Pre-infusion: number analyzed (Surgeries) | 25
  Pre-infusion | 14.0 [12.0 to 16.0]
  15 minutes post infusion: number analyzed (Participants) | 19
  15 minutes post infusion: number analyzed (Surgeries) | 23
  15 minutes post infusion | 14.0 [12.0 to 16.0]
  Change at 15 minutes post infusion: number analyzed (Participants) | 19
  Change at 15 minutes post infusion: number analyzed (Surgeries) | 23
  Change at 15 minutes post infusion | 0.0 [0.0 to 0.0]

24. Secondary Outcome: Clinically Significant Changes in Vital Signs - Pulse Rate
Description: Changes in the pulse rate (beats/minute) were assessed 15 minutes after the PK/IR infusion and compared to the pre-infusion values.
Time Frame: Vital signs measurement prior to the PK/IR infusion and 15 minutes post-infusion.
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: beats/minute
Units Other Than Participants: Surgeries
Arm/Group | BAX855
Number analyzed (Participants) | 22
Number analyzed (Surgeries) | 29
beats/minute
  Pre-infusion: number analyzed (Participants) | 20
  Pre-infusion: number analyzed (Surgeries) | 25
  Pre-infusion | 70.0 [68.0 to 74.0]
  15 minutes post infusion: number analyzed (Participants) | 19
  15 minutes post infusion: number analyzed (Surgeries) | 23
  15 minutes post infusion | 70.0 [66.0 to 77.0]
  Change at 15 minutes post infusion: number analyzed (Participants) | 19
  Change at 15 minutes post infusion: number analyzed (Surgeries) | 23
  Change at 15 minutes post infusion | -1.0 [-3.0 to 2.0]

25. Secondary Outcome: Clinically Significant Changes in Routine Laboratory Parameters- Hematology and Chemistry
Description: Changes in clinical chemistry and hematology parameters from a normal or abnormal not clinically significant (ncs) result at screening to an abnormal and clinically significant (cs) result at the end of study assessment (EOS) are listed. Changes did occur in the following laboratory parameters: Alanine Aminotransferase (ALT) (U/L), Hemoglobin (g/L), Hematocrit, Erythrocytes(TI/L), Eosinophils/Leucocytes.
Time Frame: Throughout the entire study period from screening to completion/termination (variable for each participant and depends on the nature of the invasive procedure (treatment period ranged from 43 days to 162 days).
Population: The outcome measure data include surgical enrollments with results both at screening and at the end of the study for each assay.
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Groups:
- Hemoglobin: Abnormal Ncs at Screening - Abnormal cs at EOS: Hematology: The hemoglobin result was abnormal not clinically significant at the screening assessment and changed to abnormal clinically significant at the end of study assessment.
- Hematocrit: Abnormal Ncs at Screening - Abnormal cs at EOS: Hematology: The hematocrit result was abnormal not clinically significant at the screening assessment and changed to abnormal clinically significant at the end of study assessment.
- Erythrocytes: Normal at Screening - Abnormal cs at EOS: Hematology: The Erythrocytes result was normal at the screening assessment and changed to abnormal clinically significant at the end of study assessment.
- Eosinophils/Leucocytes: Normal at Screening Abnormal cs at EOS: Hematology: The Eosinophils/Leucocytes result was normal at the screening assessment and changed to abnormal clinically significant at the end of study assessment.
- ALT: Normal at Screening - Abnormal cs at EOS: Chemistry: The ALT result was normal at the screening assessment and changed to abnormal clinically significant at the end of study assessment.
Arm/Group | Hemoglobin: Abnormal Ncs at Screening - Abnormal cs at EOS | Hematocrit: Abnormal Ncs at Screening - Abnormal cs at EOS | Erythrocytes: Normal at Screening - Abnormal cs at EOS | Eosinophils/Leucocytes: Normal at Screening Abnormal cs at EOS | ALT: Normal at Screening - Abnormal cs at EOS
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
Number analyzed (Surgeries) | 26 | 25 | 26 | 26 | 27
Surgeries | 1 | 1 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Throughout the entire study period (2 years and 9 months). For each participant the duration of treatment and therefore the entire study period depended on the nature of each participants invasive procedure (ranged from 43 days to 162 days).
Description: Adverse Events (AEs) were recorded throughout the entire study period from screening to completion/termination. AEs that occurred during or after study treatment are summarized here, AEs that occurred prior to study treatment were listed separately and are not included.
Arm/Group | BAX855
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 8/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX855 (N=22)
Device related infection (Infections and infestations) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (2)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAX855 (N=22)
Peritonsillitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication. The sponsor requires a review of results communication (e .g. for confidential information) >= 30 days prior to submission and may request an additional delay of <=180 days (e .g. for intellectual property protection).